CLINICAL TRIAL: NCT01511224
Title: A Prospective Observational Study of Patients With Drug Resistant Acinetobacter Baumannii Bacteremia Treated With Antibiotics Therapy
Brief Title: A Prospective Observational Study of Patients With Drug Resistant Acinetobacter Baumannii Bacteremia
Acronym: ANTI-AB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NTUH-TD-B-111-001
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Acinetobacter Bacteraemia
Keywords: Bloodstream infections; Acinetobacter; Drug resistant Acinetobacter baumannii bacteremia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be collected on the day of enrollment (Day 0), Day 1, 2, 3 and 7 for PCR identification and quantification of Acinetobacter species.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Colistin monotherapy
- Colistin based combination therapy: Colistin-Tigecycline, Colistin-Carbapenem, Colistin-Rifampin, Colistin-HD Unasyn
- Non-colistin containing regime
- Glycopeptide with colistin combination
- Colistin with loading dose

SUMMARY:
Extensively and multi-drug resistant A. baumannii (AB) represent an emerging threat in hospitals locally and worldwide. There is lack of prospective comparative clinical data to guide optimal strategy for treating such infections. Since it remains unclear how to treat bacteremia caused by AB, the present study aims to enroll patients at multiple sites with extensively drug resistant Acinetobacter species bacteremia receiving different combination therapy to assess treatment outcomes and analyze risk factors associated with mortality.

DETAILED DESCRIPTION:
Patients with AB bacteremia receiving antimicrobial therapy are eligible for this multicenter study. Antimicrobial agents are decided at the discretion of the attending clinical team. Clinical data to be collected include patient demographics (age, gender, underlying diseases, Pitt Bacteremia Score [20], duration of ICU stay and hospitalization before the day of first positive blood culture, central venous catheterization), antimicrobial agents on the day of bacteremia, regimens and durations of combination therapy after enrollment, and outcomes (sequential quantification change of blood A. baumannii polymerase chain reaction [PCR], survival at day 30 after enrollment, and adverse drug reactions of antimicrobial agents). Blood sample will be collected on the day of enrollment (Day 0), Day 1, 2, 3 and 7 for PCR quantification of A. baumannii and for genospecies identification. Primary end points are the interval from study enrollment to negative blood A. baumannii PCR and blood sterilization. Secondary end points are survival at 14 and 30-day after enrollment, adverse drug reactions of antimicrobial agents, and risk factors for survival at 30-day after enrollment. Inclusion criteria: 1. Adults >16 years 2. With blood culture isolate(s) A. baumannii. 3. Informed consent gained. Exclusion criteria: 1. Second/repeat episodes of bacteremia 2. Patients who could not or did not receive antimicrobial treatment 3. Patient not admitted to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adults ( >16 years)
* With blood culture isolate(s) A. baumannii
* Informed consent gained

Exclusion Criteria:

* Second/repeat episodes of bacteremia
* Patients who could not or did not receive antimicrobial treatment
* Patient not admitted to hospital

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted on intensive care units as well as general ward with AB bacteremia receiving antimicrobial therapy are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Microbiological clearance from blood | Day 0,1,2,3,7
  Interval from positive to negative blood A. baumannii PCR and blood sterilization.

SECONDARY OUTCOMES:
Survival | 14, 30, in-hospital stay
  Survival at 14, 30-day after enrollment. Survival to discharge.
Adverse drug reactions | Day 0,1,2,3,7,14
  Nephrotoxicity by RIFLE criteria
Subsequent infections and colonization | During same admission or within 1 week of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yun Sun, MD, Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - Yunlinn NTUH Branch, Douliu
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei